CLINICAL TRIAL: NCT00871975
Title: Diagnostic Utility of Tetra-NIRS in Conjunction With Urodynamic Studies
Brief Title: Tetra-NIRS Clinical Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment exceeding trial deadlines
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C001-C0015 TETRA-NIRS; NCT00849225 (obsolete NCT alias)
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder
Keywords: LUTS; OAB
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urodynamics + Tetra (Experimental): All patients were recruited to the same arm and receive Urodynamics testing as part of the routine diagnostic work-up, plus the Tetra-NIRS intervention.
  Interventions: Device: Urodynamics + TETRA - NIRS

INTERVENTIONS:
Device: Urodynamics + TETRA - NIRS — Urodynamics will be performed as per standard of care for patients enrolled, whereby one catheter is inserted into the bladder and one in the rectum to analyze bladder filling, storage and voiding conditions via pressures measured and urine flow rates detected by a uroflowmeter. Tetra-NIRS will be concurrently performed where Tetra-NIRS unit uses near infrared light at 3 different wavelengths to measure changes in haemoglobin and cytochrome. A patch is applied externally to measure these changes in the detrusor muscle of the human bladder wall. This process is similar to what is used for cerebral and muscle oxygenation monitoring (e.g., pulse oximetry). Previous clinical feasibility studies have identified a correlation between the changes in haemoglobin and cytochrome and the pressure values obtained during urodynamics procedures.

SUMMARY:
The purpose of this evaluation is to validate the previous clinical study results using a Near-Infrared Spectroscopy (NIRS) device, as compared to the conventional urodynamics (UDS) testing. The experiment will use the commercially available Tetra-NIRS and Laborie UDS equipment.

The hypothesis is that the Tetra-NIRS device, in the clinical environment, provides data to enhance the analysis using the standard urodynamics equipment (stand-alone Urodynamic procedure).

DETAILED DESCRIPTION:
This is a study of the commercially available Tetra-NIRS device to compare the results collected against conventional urodynamics. The study will evaluate male patients with lower urinary tract symptoms (LUTS) as well as female subjects with over-active bladder (OAB).

The Tetra-NIRS unit uses near infrared light at 3 different wavelengths to measure changes in haemoglobin and cytochrome from the detrusor muscle from the human bladder wall. This process is similar to what is used for cerebral and muscle oxygenation monitoring (e.g., pulse oximetry). Previous clinical feasibility studies have identified the correlation between the changes in haemoglobin and cytochrome of the bladder, and bladder pressure values obtained during urodynamics procedures and uroflow procedures.

For this study the Tetra-NIRS results will not be used by the urologist/nurse to guide in patient management and treatment decisions, but rather will only be used to collect measurements from the patient for the purposes of this study. The Tetra-NIRS sensor patch will be adhered externally to the skin surface where the bladder is located.

For this study, a minimum of 30 male subjects with LUTS and 30 female subjects with OAB scheduled to undergo a urodynamics procedure are to be enrolled. Up to 20 female subjects with OAB will be enrolled. The investigators will attempt to equally enrol male subjects into each of the two categories including obstructed and non-obstructed groups according to prostate hyperplasia (equivocal subjects will be determined by the investigator).

ELIGIBILITY:
Inclusion Criteria:

* The selection of subjects enrolled for testing must meet the following criteria:

  * Subjects must be 18 years of age or older.
  * Subjects are patients of one of the institutions and are currently scheduled for UDS
  * Male subjects must have LUTS
  * Female subjects must have OAB
  * Subjects must give their informed consent prior to enrolment.

Exclusion Criteria:

* The patient has an existing health condition which the investigators feel will not allow for safe or accurate measurements with the Tetra-NIRS device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sender Herschorn, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Vanderbilt University, Nashville, Tennessee, United States
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data are highly reliant on expert interpretation on a case-by-case basis.

REFERENCES:
- [Result] Mastoroudes H, Giarenis I, Vella M, Srikrishna S, Robinson D, Cardozo L, Karrouze I, Campbell A, Macnab A. Use of near infrared spectroscopy as an alternative to videourodynamics to detect detrusor overactivity in women with the overactive bladder syndrome. Urology. 2012 Sep;80(3):547-50. doi: 10.1016/j.urology.2012.05.036. Epub 2012 Jul 26. PMID 22840868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each site recruited in a Urology clinic setting. All patients were scheduled for Urodynamics testing. Sunnybrook recruitment period spanned Apr 2010 - Feb 2012. Vanderbilt Sept 2009 - May 24 2010. King's College May 2010 - August 2010.
Pre-assignment Details: There were no group assignments.
Groups:
- Urodynamics + Tetra-NIRS: Single arm - all patients were recruited following a requirement for urodynamic testing. The patient is the invited to the clinic room to perform the urodynamics test concurrently with the Tetra-NIRS device. The clinic staff perform urodynamics per their standard protocol, with the Tetra-NIRS patch applied externally above the location of the bladder. The numerical pressure data resulting from the urodynamics machine plus the hemoglobin levels (oxygenated and deoxygenated) measured by the Tetra-NIRS device are displayed on a computer and saved. The test would take approx. 45 minutes to perform, after which time the patient is free to go home. Interpretation of the Tetra-NIRS had no bearing on the patients' diagnosis, however urodynamic interpretation was performed per their standard protocol.
Period: Overall Study
Arm/Group | Urodynamics + Tetra-NIRS
Started | 155
Completed | 133
Not Completed | 22
Not completed — Technical difficulty w155-1ith equipment | 3
Not completed — Catheters could not be inserted | 1
Not completed — Patient unable to void/insufficient vol | 13
Not completed — Motion artifact, tracing uninterpretable | 5

BASELINE CHARACTERISTICS:
Population: Includes both male patients suffering from LUTS, and female patients suffering from OAB.
Arm/Group | Urodynamics + Tetra-NIRS
Number analyzed (Participants) | 155
Age, Customized [Number; unit: participants]
  Greater than or equal to 18 years | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 18
  Canada | 37
  United Kingdom | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urodynamic Detrusor Overactivity Events or Prostatic Obstruction as Detected by Tetra-NIRS Compared to Urodynamics
Description: The Tetra-NIRS device provides a linear pattern similar to the pressures obtained during urodynamics. The NIRS output shows relative change in hemoglobin concentrations (oxygenated and deoxygenated) where the numerical value does not actually indicate the concentration, so there is no unit of measure. The numerical output is used to track change over time, or trendline analysis. A qualified interpreter studied tracings for significant changes (+/-2 Hb units) in the NIRS patterning during detrusor overactivity events. As well, under its' approved intended use, Tetra-NIRS trendline analysis was compared against urodynamics during voiding in males, such that a downward trend during voiding indicates urethral obstruction, and an upward trend indicates an unobstructed urethra.
Time Frame: 1 Year
Population: Male and female patients were included, where the urodynamics tracings were compared against the Tetra NIRS tracings.
Measure: Number; unit: participants
Groups:
- Urodynamics + Tetra NIRS: Single arm - all patients were recruited following a requirement for urodynamic testing. The patient is the invited to the clinic room to perform the urodynamics test concurrently with the Tetra-NIRS device. The clinic staff perform urodynamics per their standard protocol, with the Tetra-NIRS patch applied externally above the location of the bladder. The numerical pressure data resulting from the urodynamics machine plus the hemoglobin levels (oxygenated and deoxygenated) measured by the Tetra-NIRS device are displayed on a computer and saved. The test would take approx. 45 minutes to perform, after which time the patient is free to go home. Interpretation of the Tetra-NIRS had no bearing on the patients' diagnosis, however urodynamic interpretation was performed per their standard protocol.
Arm/Group | Urodynamics + Tetra NIRS
Number analyzed (Participants) | 133
participants
  True Positive on Tetra-NIRS + UDS | 30
  False Positive on Tetra-NIRS + UDS | 59
  False Negative on Tetra-NIRS + UDS | 10
  True Negatives on Tetra-NIRS + UDS | 34
Statistical Analysis 1: Comparison: Urodynamics + Tetra NIRS; A contingency table was used to compare presence or absence of an event (eg. detrusor overactivity) on the urodynamic tracing with interpretation of events on the Tetra-NIRS tracings; Test type: Superiority or Other; Sensitivity (percent) = 80.6 — We found an 80.6% sensitivity for detection of detrusor overactivity on Tetra-NIRS as compared to urodynamics
Statistical Analysis 2: Comparison: Urodynamics + Tetra NIRS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Specificity (percent) = 28.1 — We found a 28.1% specificity for detection of detrusor overactivity on Tetra-NIRS as compared to urodynamics

ADVERSE EVENTS:
Arm/Group | Urodynamics + Tetra-NIRS
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

LIMITATIONS AND CAVEATS:
Early termination was due to slow recruitment exceeding trial deadlines. Technical issues resulted in several studies being excluded (8).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No